CLINICAL TRIAL: NCT01475123
Title: Effects of Nicorandil on Cardiovascular Events in Patients With Coronary Artery Disease Receiving Hemodialysis
Brief Title: Prospective Study of End Stage Renal Disease Patients With Coronary Artery Disease Treated by Oral Nicorandil
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Yasuhiro Nagayoshi, principal investigator, Kumamoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVM-2008-PRECON
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; End Stage Renal Disease
Keywords: Nicorandil; Randomized control study; Hemodialysis; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Kidney Failure, Chronic | interventions — Nicorandil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicorandil (Active Comparator): Nicorandil was administered orally (15mg/day).
  Interventions: Drug: Nicorandil
- Non-nicorandil (No Intervention): Nicorandil was not administered.

INTERVENTIONS:
Drug: Nicorandil — 15mg per day
  Other Names: Sigmart
  Arms: Nicorandil

SUMMARY:
Nicorandil is potentially effective to prevent cardiovascular events in patients with coronary artery disease (CAD) receiving hemodialysis. The purpose of this study is to prospectively investigate whether nicorandil is effective in reducing the incidence of cardiovascular events in patients with CAD on hemodialysis.

DETAILED DESCRIPTION:
Patients on hemodialysis for end-stage renal disease are at high risk for death from ischemic heart disease. It was reported that nicorandil, a hybrid compound on adenosine triphosphate-sensitive potassium channel opener and nitric oxide door, was potentially effective to prevent cardiovascular events in patients with CAD receiving hemodialysis. Therefore, investigators prospectively examine whether nicorandil is effective in reducing the incidence of cardiovascular events in patients with CAD on hemodialysis.

The primary endpoint is a composite of cardiovascular death, sudden cardiac death, nonfatal myocardial infarction, hospitalization for recurrent symptomatic myocardial ischemia and stroke. The secondary endpoints are total mortality, revascularization therapy, hospitalization for heart failure, hospitalization for peripheral artery disease and newly onset of atrial fibrillation.

Patient population that needs to prove the hypothesis is estimate to be 300 cases in total (150 cases in each group). Investigators set the parameters which are need to calculate the number of study patients as follows; drop out rate 10%, an event rate of the primary end point for two years 50%, a risk reduction rate brought by nicorandil 60%, a statistical power 80% and two-sided significant level 0.05. Investigators referred the event rate and the risk reduction rate from the previous study by Ishi H et al. In this study, event rate of the primary end point for two years was 50% and the risk reduction brought by nicorandil was 60%. Event rate of the present study will be lower, because drug-eluting stents are widely used to prevent restenosis in the present era. Moreover, investigators include the patients underwent coronary bypass graft in the present study. In addition, non-cardiovascular mortality is high in the patients on hemodialysis. Considering all the various factors together, investigators estimated the study sample size.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients are who meet the following criteria:

* Patient with previously diagnosed coronary artery disease (significant coronary artery stenosis is defined as > 75% narrowing of the artery lumen)
* Patients who continued hemodialysis for more than one month

Exclusion Criteria:

* Within one month after acute myocardial infarction
* Within 3 months after coronary artery bypass graft (CABG)
* Treatment with phosphodiesterase type 5 inhibitor
* Candidates for carotid artery stenting
* Severe disease requiring active medical treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is composite of :1) cardiovascular death 2)sudden cardiac death 3)nonfatal myocardial infarction 4)Hospitalization for recurrent symptomatic myocardial ischemia 5)stroke | 2 years

SECONDARY OUTCOMES:
Total mortality | 2 years
revascularization therapy | 2 years
hospitalization for heart failure | 2 years
hospitalization for peripheral artery disease | 2 years
newly onset of atrial fibrillation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, MD, PhD, Study Chair — Kumamoto University
Locations (1):
- Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University, Kumamoto, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ishii H, Toriyama T, Aoyama T, Takahashi H, Yamada S, Kasuga H, Ichimiya S, Kanashiro M, Mitsuhashi H, Maruyama S, Matsuo S, Naruse K, Matsubara T, Murohara T. Efficacy of oral nicorandil in patients with end-stage renal disease: a retrospective chart review after coronary angioplasty in Japanese patients receiving hemodialysis. Clin Ther. 2007 Jan;29(1):110-22. doi: 10.1016/j.clinthera.2007.12.020. PMID 17379051